CLINICAL TRIAL: NCT03191565
Title: The mDIARY Study: Using Smartphones for Daily Selfmonitoring of Skilluse and Outcome in Dialectical Behavior Therapy With Borderline Personality Disorder: A Combined RCT and Timeseries Study
Brief Title: Using Smartphones for Selfmonitoring of Skill-use i Dialectical Behavior Therapy
Acronym: mDIARY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other); Innovation Fund Denmark (Individual); Monsenso (Industry); Mclean Hospital (Other); Central Denmark Region (Other)
Responsible Party: Principal Investigator, Stig Helweg-Jørgensen, Principal investigator, Region of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDUSF-20216-56-(556)
Record Dates: First submitted 2017-03-24; First posted 2017-06-19 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Borderline Personality Disorder; Emotional Instability; Skill, Coping
Keywords: mhealth; self-monitoring; Outcome monitoring
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-Condition (Experimental): In this condition the intervention is that participants enter their skills-use and mood on a smartphone. They can follow their progress on graphs on the smartphone, get reminders to train skills, get psychoeducation about what the different emotion regulation coping skills can do, and how to do the skills. therapists can watch patient progress online, and review skill use together with the patients while in psychotherapy. The intervention is using a smartphone as an adjunct to the treatment.
  Interventions: Device: Monsenso DBT-app and IT monitoring program
- Paperdiary-condition (Active Comparator): Patients are, weekly, given a paper diary sheet to fill out on a daily basis at home No prompting, no accumulative overview of progress. Patients are supposed to bring this paper to the weekly therapysession
  Interventions: Other: Paper diary sheet

INTERVENTIONS:
Other: Paper diary sheet — Writing skill-use and symptoms on a week matrix type sheet
  Arms: Paperdiary-condition
Device: Monsenso DBT-app and IT monitoring program — Entering skill-use and symptoms on a smartphone with Monsenso DBT-app and IT monitoring program
  Arms: App-Condition

SUMMARY:
BACKGROUND: Borderline Personality Disorder (BPD) is a serious and debilitating mental disease characterized by difficulties with emotion regulation that leads to unstable and self- destructive behavior and relationships. The prevalence of BPD is between 1% and 5% in the Scandinavian population with similar prevalence rates found in US epidemiologic surveys. BPD increases the risk for suicide by 4-fold, while patients with comorbid BDP and tendency to self-harm have a further 2-fold attenuated risk. BDP is difficult to treat, and even more difficult when co-occurring with other disorders. Dialectical Behavior Therapy (DBT) is the best validated treatment for BPD, showing medium to large effect sizes as compared to treatment as usual for anger, parasuicidality (suicide attempts without an intention to die) and poor mental health. DBT uses self-monitoring as the mainstay of treatment, which helps patients regulate their emotions by means of emotional regulating skills, and reduce problem behavior. Self-monitoring has traditionally been done by means of daily paper diaries. The latest developments in smartphone applications have generated alternatives for ecological momentary assessments of problematic behavior that even prompt patients to practice skills targeting emotion regulation. An example of this is Monsenso's DBT self-monitoring mHealth application (mHealth means mobile health, public health supported by mobile phones). Such applications may enhance treatment success in BPD patients, as they are available to patients at all times.

OBJECTIVES: To evaluate the Monsenso's mHealth app with respect to clinical efficacy as an adjunct to DBT-psychotherapy treatment and utility as a way to measure outcomes in BPD patients.

METHODS: The study will be a 2-year multi center, randomized controlled trial. In both conditions patients will be followed for one year. Self report data of DBT-skills-use, positive and negative affect, Standardised self report questionnaires on Emotion regulation ability; functioning; borderline symptoms. will be given pre, post and every month. The treatment arm (n=50) will receive the mHealth app that includes coaching suggestions and instructed how to use it. The control arm (n=50) will only use a pen and paper based self-monitoring, as traditionally used in DBT-treatment.

STUDY ENDPOINTS: Primary: mean number of days passed per new DBT-Skill learned. Secondary: Borderline personality disorder(BPD)-symptoms, Emotion regulation ability, ratio positive/negative affect.

DETAILED DESCRIPTION:
BACKGROUND

Borderline personality disorder

It is estimated that 1-5% of the Scandinavian population meets the criteria for borderline personality disorder (BPD). General consensus regarding estimates for the western world population, is that around 1,5% of the population meets criteria for BPD. Lifetime prevalence will be estimated as 3 times as high (about 5%). The percentage for clinical populations is considerably higher and is estimated to be around 28% (range 9.3 to 46.3 % of patients in different current studies) of all psychiatric patients meeting this diagnosis. BDP is characterized by an instability across a number of domains: Mood, interpersonal relationships, self-image, impulse- and behavioral control. Generally, these BDP manifestations are attributed to a lack of ability to emotionally regulate. Patients with BDP have a four times increased risk of premature death compared to the general population, emphasizing the need for appropriate treatment.

Treatment of borderline personality disorder

Dialectical behavior therapy (DBT) has shown good clinical efficacy and is regarded as one of the most well researched evidence-based treatments for BPD. The DBT treatment centers around the learning of a predefined set of behavioral skills, targeting lack of emotional, mental and behavioral self-control. These skills are trained in group and individual therapy.

In standard clinical practice, evaluation of a patient's progress in learning skills is left to the clinician's subjective memory and evaluation of weekly data.

Self-monitoring of skill use and accompanying changes in suicidality, self-harm, and emotional reactivity have traditionally been done by means of paper diaries. Technological advances in self-monitoring might reduce the burden on the patient, increase data quality and generate new opportunities for registration (8). Recent studies on pain management have suggested that mhealth solutions significantly increase compliance. Studies using electronic diaries in the treatment of bipolar disorders, in pain- and weight management, and in patients treated with chemo-therapy have also shown promising results. DBT skills have been shown to mediate improvements in BPD defining behaviors.

However, no randomized studies to date have examined if a mobile phone-/mhealth solution could speed up the time it takes for patients to assimilate the DBT-skills, while at the same time serving the function of filling out diary cards for the treatment of BDP.

Regarding the time series part of the study, a single pilot study of ecological momentary assessment (EMA) has demonstrated significant differences in fluctuations of positive and negative affect on a daily basis when comparing major depressive disorder to BPD. Hence, this lends promise that a purpose-designed mobile phone application aimed at collecting DBT-diary data will produce time-efficient and valid data of higher quality than traditional paper-registrations. This will also at the same time generate objective outcome data, thus collecting multimodal data. Both self report and passive sensor data. The exact same sensor data have been shown to have value in predicting manic episodes in bipolar patients.

When starting an mhealth-supported session, it is possible to view the EMA data (for content, see Table 1), self-rated daily assessments, monthly questionnaires together with the therapist. The mDiary system will automatically generate chosen relevant questionnaires at a selected ratio, making the research data-collection much easier. The patient and the therapist can also get access to phone sensor data, such as activity level, phone use, internet use and minutes of communication on phone as well.

The increased overview provided by diarycard-, sensor- and questionnaire data can also be useful when evaluating and discussing patient cases at staff meetings or during therapist supervision.

ELIGIBILITY:
Inclusion Criteria:

* Must be admitted to DBT treatment at a psychiatric hospital treatment facility in Denmark
* Must meet the criteria for Emotionally unstable personality disorder
* Must be 18 yr.o.

Exclusion Criteria:

* Psychosis
* Schizophrenia
* Bipolar disorder
* IQ under 70
* Patients who do not have a working smartphone
* Demographic data on rejected patients will be collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Days/skill | Daily measurements up to 1 year. (minimum 8 months.)
  Mean number of days required to learn a new DBT-skill

SECONDARY OUTCOMES:
Borderline symptoms | Pre, post and monthly measurements up to 1 year (minimum 8 months)
  BPD symptoms according to the ZAN-BPD
Ability to emotionally regulate | Pre, post and monthly measurements up to 1 year (Minimum 8 months)
  Emotion regulation ability according to the Kim Gratz DERS-scale
Compliance to self registration | Daily measurements up to 1 year (minimum 8 months)
  Days of compliant registration

CONTACTS AND LOCATIONS:
Overall Officials: Stig Helweg-Jørgensen, PsyD, Principal Investigator — Region of Southern Denmark
Locations (5):
- Denmark (5):
  - Glostrup DAT team. Psykiatrisk Ambulatorium, Copenhagen, Brøndby
  - Haderslev DAT team, Haderslev
  - Silkeborg DAT team, Psykiatriens Hus, Silkeborg
  - Lokalpsykiatrisk ambulatorium, Svendborg
  - Vejle DAT- team, Psykiatrisk ambulatorium, Vejle

IPD SHARING:
Plan to Share IPD: Yes
After receiving permission from the participants, individual data will be shared with the individual therapist who is treating the patient, but only data regarding for their own clients, so they can follow therapy-progress. De-identified data will be shared with researcher doing the economic evaluation, August 2019. According to danish data protection law this researcher will need a Data processor approval through The danish Data protection agency.

REFERENCES:
- [Background] Torgersen S, Kringlen E, Cramer V. The prevalence of personality disorders in a community sample. Arch Gen Psychiatry. 2001 Jun;58(6):590-6. doi: 10.1001/archpsyc.58.6.590. PMID 11386989
- [Background] Torgersen S. [Paranoid schizophrenia, paranoid psychoses and personality disorders]. Tidsskr Nor Laegeforen. 2012 Apr 17;132(7):851-2. doi: 10.4045/tidsskr.12.0318. No abstract available. Norwegian. PMID 22511105
- [Background] Stoffers JM, Vollm BA, Rucker G, Timmer A, Huband N, Lieb K. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD005652. doi: 10.1002/14651858.CD005652.pub2. PMID 22895952
- [Background] Stone AA, Broderick JE, Schwartz JE, Shiffman S, Litcher-Kelly L, Calvanese P. Intensive momentary reporting of pain with an electronic diary: reactivity, compliance, and patient satisfaction. Pain. 2003 Jul;104(1-2):343-51. doi: 10.1016/s0304-3959(03)00040-x. PMID 12855344
- [Background] Faurholt-Jepsen M, Vinberg M, Frost M, Christensen EM, Bardram JE, Kessing LV. Smartphone data as an electronic biomarker of illness activity in bipolar disorder. Bipolar Disord. 2015 Nov;17(7):715-28. doi: 10.1111/bdi.12332. Epub 2015 Sep 23. PMID 26395972
- [Background] Turk MW, Elci OU, Wang J, Sereika SM, Ewing LJ, Acharya SD, Glanz K, Burke LE. Self-monitoring as a mediator of weight loss in the SMART randomized clinical trial. Int J Behav Med. 2013 Dec;20(4):556-61. doi: 10.1007/s12529-012-9259-9. PMID 22936524
- [Background] Burke LE, Styn MA, Sereika SM, Conroy MB, Ye L, Glanz K, Sevick MA, Ewing LJ. Using mHealth technology to enhance self-monitoring for weight loss: a randomized trial. Am J Prev Med. 2012 Jul;43(1):20-6. doi: 10.1016/j.amepre.2012.03.016. PMID 22704741
- [Background] Faurholt-Jepsen M, Frost M, Ritz C, Christensen EM, Jacoby AS, Mikkelsen RL, Knorr U, Bardram JE, Vinberg M, Kessing LV. Daily electronic self-monitoring in bipolar disorder using smartphones - the MONARCA I trial: a randomized, placebo-controlled, single-blind, parallel group trial. Psychol Med. 2015 Oct;45(13):2691-704. doi: 10.1017/S0033291715000410. Epub 2015 Jul 29. PMID 26220802
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Neacsiu AD, Eberle JW, Kramer R, Wiesmann T, Linehan MM. Dialectical behavior therapy skills for transdiagnostic emotion dysregulation: a pilot randomized controlled trial. Behav Res Ther. 2014 Aug;59:40-51. doi: 10.1016/j.brat.2014.05.005. Epub 2014 May 27. PMID 24974307
- [Background] Bedics JD, Atkins DC, Comtois KA, Linehan MM. Weekly therapist ratings of the therapeutic relationship and patient introject during the course of dialectical behavioral therapy for the treatment of borderline personality disorder. Psychotherapy (Chic). 2012 Jun;49(2):231-40. doi: 10.1037/a0028254. PMID 22642526
- [Background] Klein AS, Skinner JB, Hawley KM. Targeting binge eating through components of dialectical behavior therapy: preliminary outcomes for individually supported diary card self-monitoring versus group-based DBT. Psychotherapy (Chic). 2013 Dec;50(4):543-52. doi: 10.1037/a0033130. PMID 24295464
- [Derived] Laursen SL, Helweg-Jorgensen S, Langergaard A, Sondergaard J, Sorensen SS, Mathiasen K, Lichtenstein MB, Ehlers LH. Mobile Diary App Versus Paper-Based Diary Cards for Patients With Borderline Personality Disorder: Economic Evaluation. J Med Internet Res. 2021 Nov 11;23(11):e28874. doi: 10.2196/28874. PMID 34762057
- [Derived] Helweg-Jorgensen S, Beck Lichtenstein M, Fruzzetti AE, Moller Dahl C, Pedersen SS. Daily Self-Monitoring of Symptoms and Skills Learning in Patients With Borderline Personality Disorder Through a Mobile Phone App: Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2020 May 25;9(5):e17737. doi: 10.2196/17737. PMID 32449690
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793